CLINICAL TRIAL: NCT03598881
Title: A Study to Assess the Impact of a Non-SLS Toothpaste Upon Oral Mucosal Desquamation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Collaborators: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: ORL-OSS-2545
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Sloughing Skin; Mucosal Inflammation
MeSH Terms: conditions — Necrosis; Mucositis | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Toothpaste containing 0.32%NaF and no sodium lauryl sulphate (SLS)
  Interventions: Other: Treatment
- Comparator (Active Comparator): Toothpaste containing 0.8% sodium monofluorophosphate (SMFP) and sodium lauryl sulphate (SLS)
  Interventions: Other: Treatment

INTERVENTIONS:
Other: Treatment

SUMMARY:
This study is to compare the effect on oral mucosal desquamation of a non-SLS toothpaste and an SLS-containing toothpaste..

DETAILED DESCRIPTION:
Subjects will use a wash out toothpaste for at least 10 days prior to each leg of the crossover design. Clinical assessment of oral mucosa status will be performed by a trained examiner before supervised product application, 30 minutes after product application and again after 4 days of twice daily brushing with product. Supervised product application consists of cap splint application of allocated toothpaste to maxillary arch followed by brushing whole mouth with toothpaste and swishing with resultant slurry around the mouth.

For visual sloughing evaluation, the oral mucosa will be divided into 12 assessment areas and each area evaluated for severity of sloughing on a 0 to 5 scale.

The following outcomes will be generated from the sloughing data:

1. Whole mouth data per subject: each non-zero severity score will be treated as one lesion count, giving a maximum score of 12;
2. Subject level mucosal severity sloughing score: severity score averaged over the 12 areas assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Internal (University of Birmingham Dental School) panellists only
2. Willing to sign an informed consent form and complete a medical history questionnaire.
3. Must be available for the duration of the study.
4. Must be a current non-smoker and not chew tobacco.
5. Have a minimum of 8 teeth in both upper and lower jaws, which are free from obvious untreated caries or significant periodontal disease

Exclusion Criteria:

1. Show unwillingness, inability or lack of motivation to carry out the study procedures
2. Are pregnant or breastfeeding females.
3. Are diabetic.
4. Have severe oral mucosal problems.
5. Orthodontic banding or removable partial dentures
6. Have an active cold sore.
7. Have any oral piercings.
8. Have a mouth ulcer or who experience mouth ulcers on a regular basis, Lichen Planus Vesiculo-Bullous disorders
9. Obvious signs of untreated caries or significant periodontal disease, which in the opinion of the Study Dentist, will effect either the scientific validity of the study or if the volunteer's participation would affect their well being
10. Volunteers who are at risk from transient bacteraemias.
11. Regular use of medication, which could interfere with study objectives or affect the validity of the study.
12. Have or have had a medical or dental condition, which in the option of the dentist would make them unsuitable for inclusion.
13. Have problem of bleeding after brushing.
14. Must not be a regular user of chlorhexidine mouthwash, or have used it within the past 6 weeks.
15. Has allergic responses to dental/oral hygiene products or components in the formulation of the toothpaste.
16. The subject is participating in other studies testing oral care products.
17. The subject is an employee of Unilever.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-09-19 (Actual); Primary Completion 2016-11-21 (Actual); Study Completion 2016-11-21 (Actual)

PRIMARY OUTCOMES:
Aggregate number of lesions | 30 minutes
  Total lesion count aggregated across all subjects
Aggregate number of lesions | 4 days
  Total lesion count aggregated across all subjects

SECONDARY OUTCOMES:
Lesion severity | 30 minutes
  Subject level mucosal severity sloughing score
Lesion severity | 4 days
  Subject level mucosal severity sloughing score

CONTACTS AND LOCATIONS:
Overall Officials: Iain Chapple, Professor, Principal Investigator — The University of Birmingham
Locations (1):
- University of Birmingham, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No